CLINICAL TRIAL: NCT05356065
Title: The Turkish Version of the Oslo Sports Trauma Research Center (OSTRC) Questionnaire on Overuse Injuries and Health Problems; Validity and Reliability Study
Brief Title: The Turkish Version of the OSTRC Questionnaires
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şeyda ÖZAL, Principal Investigator (Master of Science degree Physiotherapist), Gazi University
Other Study IDs: GAZIUN
Record Dates: First submitted 2022-04-14; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Sports Injury
Keywords: overuse injury; athlete health; outcome measures; validity and reliability study
MeSH Terms: conditions — Athletic Injuries; Cumulative Trauma Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey administration — Outcome Measures

SUMMARY:
Exposure to repetitive activities and heavy workloads makes athletes vulnerable to overuse injuries over time. Well-timed detection of these injuries is crucial to maintaining their sports career healthily. The Oslo Sports Trauma Research Centre questionnaires for Overuse Injury (OSTRC-O) and Health Problems (OSTRC-H) are universally used as valid and reliable tools in athlete health screening. This study aims to make them available for Turkish athletes.

The internal consistency, reproducibility, and validity of the questionnaires were analyzed. Data were obtained from 72 athletes from different sports types. 33 participants were screened weekly for six weeks to detect score changes and calculate effect sizes. Participants filled out the OSTRC-O, the OSTRC-H, the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ), and the Nottingham Health Profile (NHP) for validity analyses. The internal consistency and test-retest reliability values were very high for both questionnaires. There was a moderate correlation between OSTRC-O and OSTRC-H scores with CMDQ and NHP. The area under the curve (AUC) values were adequate for all scales. The effect size values were moderate for all scales. Turkish versions of the OSTRC-O and OSTRC-H questionnaires are valid and reliable tools for Turkish-speaking athletes in different sports branches.

DETAILED DESCRIPTION:
Introduction and Aims All athletes are vulnerable to acute traumas or cumulative injuries throughout their sports life. Thus, screening the health levels of athletes and investigating whether they have overuse injuries is essential both to prevent acute traumas and improve health and performance. There is no valid and reliable subjective measurement tool to perform this screening in athletes in Turkish currently. However, the valid and reliable "Oslo Sports Trauma Research Centre Overuse Injury Questionnaire - (OSTRC)" questionnaires are available in English. So the investigators aimed to adapt the OSTRC- Overuse (OSTRC-O) and the OSTRC-Health Questionnaire (OSTRC-H) into Turkish.

Methods Permission was obtained from the developer authors. Then, ethical approval was acquired from the clinical researches ethics committee. Questionnaires were adapted into Turkish systematically. A pilot study was conducted to ensure the accuracy of meaning and comprehensibility of translated questionnaires. Next, the validity and reliability of the new tools were estimated. 72 athletes aged between 18 and 35, who can understand and speak Turkish fluently from various sports branches, were included. Informed consent was obtained from all athletes. The demographics of the participants were recorded. All participants were administered the Cornell Musculoskeletal Discomfort Questionnaire (CMDQ), Nottingham Health Profile (NHP), OSTRC-O, and OSTRC-H questionnaires. The OSTRC-O OSTRC-H and CMDQ questionnaires were repeated weekly for six weeks on 33 athletes.

Reliability was analyzed by internal consistency and test-retest methods. The validity of the scale was evaluated in terms of content validity and concurrent validity. Content validity was verified with reports of participants at the end of the sixth week. To evaluate the concurrent validity, total OSTRC scores were compared with the total scores of CMDQ and NHP. Correlations of the OSTRC-O and OSTRC-H change scores with CMDQ change scores separately were assessed throughout the six weeks in point of the Effect Size (ES) for responsiveness. Receiver Operating Characteristic (ROC) Curve test based on the area under the curve (AUC) depicted to define the performance of these assessment tools. Statistical analyses were performed with the Statistical Package for Social Sciences Program.

ELIGIBILITY:
Inclusion Criteria:

* accepting to participate in the study
* Participating in sports

Exclusion Criteria:

* Being illiterate
* Being younger than 18 years or older than 35 years

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Athletes aged between 18 and 35, who can understand and speak Turkish fluently from various sports branches
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Oslo Sports Trauma Research Centre Questionnaires for Overuse Injury (OSTRC-O) | Baseline
  The "Oslo Sports Trauma Research Centre Questionnaires for Overuse Injury" is a self-reported outcome measure. It queries sports participation, training volume, sports performance, and pain for a selected body location-e.g. knee taking into account the last seven days. A severity score is between 0-100 points. Higher points show worse health conditions.
Oslo Sports Trauma Research Centre questionnaires on Health Problems (OSTRC-H) | Baseline
  "Oslo Sports Trauma Research Centre questionnaires on Health Problems" is a self-reported outcome measure. It is applied to determine the effects of general health problems on sports participation, training volume, sports performance, and pain for the last seven days. A severity score is between 0 and 100 points. Higher points show worse health conditions.
Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) | Baseline
  Cornell Musculoskeletal Discomfort Questionnaire is used to ascertain the musculoskeletal problems experienced in the last week during work life. Participants marked the frequency, discomfort, and interference categories for 20 different regions on the body map diagram. The total score of the questionnaire is between 0 (best condition) and 90 (worst health status).
Nottingham Health Profile (NHP) | Baseline
  Nottingham Health Profile is a self-reported outcome measure. It is a general health questionnaire consisting of 6 sub-parameters (pain, physical mobility, emotional reactions, sleep, energy level, social isolation) and 38 items. Participants marked yes or no for each item. The total score ranges from 0 to 600, and the total score is inversely proportional to the quality of life.

SECONDARY OUTCOMES:
Oslo Sports Trauma Research Centre Questionnaires for Overuse Injury (OSTRC-O) | Change from baseline score at 6 weeks
  The "Oslo Sports Trauma Research Centre Questionnaires for Overuse Injury" is a self-reported outcome measure. It queries sports participation, training volume, sports performance, and pain for a selected body location-e.g. knee taking into account the last seven days. A severity score is between 0-100 points. Higher points show worse health conditions
Oslo Sports Trauma Research Centre questionnaires on Health Problems (OSTRC-H) | Change from baseline score at 6 weeks
  "Oslo Sports Trauma Research Centre questionnaires on Health Problems" is a self-reported outcome measure. It is applied to determine the effects of general health problems on sports participation, training volume, sports performance, and pain for the last seven days. A severity score is between 0 and 100 points. Higher points show worse health conditions.
Cornell Musculoskeletal Discomfort Questionnaire (CMDQ) | Change from baseline score at 6 weeks
  Cornell Musculoskeletal Discomfort Questionnaire is used to ascertain the musculoskeletal problems experienced in the last week during work life. Participants marked the frequency, discomfort, and interference categories for 20 different regions on the body map diagram. The total score of the questionnaire is between 0 (best condition) and 90 (worst health status).

CONTACTS AND LOCATIONS:
Overall Officials: Şeyda ÖZAL, Ph.D. (c), Principal Investigator — Gazi University Faculty of Health Sciences; Nihan KAFA, Asoc. Prof., Study Director — Gazi University Faculty of Health Sciences; Fuat YUKSEL, Ph.D. (c), Principal Investigator — Gazi University Faculty of Health Sciences; Nevin A GÜZEL, Prof. Dr., Study Chair — Gazi University Faculty of Health Sciences
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It can be shared with reasonable requirements

REFERENCES:
- [Background] Bahr R, Bahr IA. Incidence of acute volleyball injuries: a prospective cohort study of injury mechanisms and risk factors. Scand J Med Sci Sports. 1997 Jun;7(3):166-71. doi: 10.1111/j.1600-0838.1997.tb00134.x. PMID 9200321
- [Background] Clarsen B, Ronsen O, Myklebust G, Florenes TW, Bahr R. The Oslo Sports Trauma Research Center questionnaire on health problems: a new approach to prospective monitoring of illness and injury in elite athletes. Br J Sports Med. 2014 May;48(9):754-60. doi: 10.1136/bjsports-2012-092087. Epub 2013 Feb 21. PMID 23429267
- [Background] Clarsen B, Myklebust G, Bahr R. Development and validation of a new method for the registration of overuse injuries in sports injury epidemiology: the Oslo Sports Trauma Research Centre (OSTRC) overuse injury questionnaire. Br J Sports Med. 2013 May;47(8):495-502. doi: 10.1136/bjsports-2012-091524. Epub 2012 Oct 4. PMID 23038786
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] Hunt SM, McKenna SP, McEwen J, Williams J, Papp E. The Nottingham Health Profile: subjective health status and medical consultations. Soc Sci Med A. 1981 May;15(3 Pt 1):221-9. doi: 10.1016/0271-7123(81)90005-5. No abstract available. PMID 6973203
- [Background] Erdinc O, Hot K, Ozkaya M. Turkish version of the Cornell Musculoskeletal Discomfort Questionnaire: cross-cultural adaptation and validation. Work. 2011;39(3):251-60. doi: 10.3233/WOR-2011-1173. PMID 21709361